CLINICAL TRIAL: NCT04014088
Title: A Randomized Controlled Trial Comparing Helmet Continuous Positive Airway Pressure (CPAP) vs Facemask CPAP for Treatment of Acute Cardiogenic Pulmonary Edema In The Emergency Department
Brief Title: Helmet CPAP vs Facemask CPAP in ACPE (hCPAP vs fCPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Raja Permaisuri Bainun (Other Government)
Responsible Party: Principal Investigator, Dr. Adi Bin Osman, Emergency Medicine Consultant, Hospital Raja Permaisuri Bainun
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-14-1894-21782 (IIR).
Record Dates: First submitted 2019-07-04; First posted 2019-07-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acute Cardiogenic Pulmonary Edema
Keywords: helmet CPAP; facemask CPAP; pulmonary edema; non invasive ventilation
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- helmet CPAP (Active Comparator): helmet CPAP administer to patient diagnosed as acute cardiogenic pulmonary edema
  Interventions: Device: hCPAP vs fCPAP
- facemask CPAP (Active Comparator): facemask CPAP administer to patient diagnosed as acute cardiogenic pulmonary edema
  Interventions: Device: hCPAP vs fCPAP

INTERVENTIONS:
Device: hCPAP vs fCPAP — The patient presented with Acute Cardiogenic Pulmonary Edema will be randomized into either helmet CPAP or facemask CPAP.

SUMMARY:
This study objectively held to compare the physiological outcomes in the non-invasive (NIV) treatment of Acute Cardiogenic Pulmonary Edema (ACPE) patients in the Emergency Department (ED) delivered by helmet CPAP (hCPAP) and facemask CPAP (fCPAP).Patients will be randomized to receive either hCPAP or fCPAP.

DETAILED DESCRIPTION:
Non-invasive ventilation(NIV) has different types of interfaces that had been used in acute cardiogenic pulmonary edema. The appropriate interface is necessary to provide comfort and lead to the success of NIV.

NIV delivered via facemask had been used widely. However, it was associated with leaks and discomfort to the patient.

Helmet continuous positive airway pressure (hCPAP) is an NIV interface that allows the provision of high airway pressures with a minimal leak.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged more than 18 years old presented with acute cardiogenic pulmonary oedema

Exclusion Criteria:

1. Age less than 18 years old
2. Low GCS (less than 8), altered mental status
3. Hemodynamic instability, impending cardiopulmonary arrest
4. Use of vasopressors, inotropes
5. Exacerbation of asthma or chronic respiratory failure
6. Urgent need for endotracheal intubation
7. Absence of airway protective gag reflex
8. Elevated intracranial pressure
9. Tracheostomy
10. Pregnant
11. Upper airway obstruction
12. Injuries or surgery to head and neck less than 6 months upon presentation
13. Claustrophobia
14. Blind or poor vision
15. Medico-legal related cases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate | 1 hour
  Respiratory rate change post intervention

SECONDARY OUTCOMES:
Heart Rate | 1 hour
  Heart rate change post intervention
Partial Pressure of Arterial Oxygen Level | 1 hour
  Partial arterial oxygen level post intervention
Ratio Of Partial Pressure Arterial Oxygen And Fraction Of Oxygen | 1 hour
  Partial arterial oxygen/fraction of oxygen ratio change post intervention
Dyspnea Scale | 1 hour
  Dyspnea scale improvement post intervention.Dyspnea scale measured using an unmarked 100mm VAS card that had mark with "I can breathe normally", at one end correspond to patients' normal baseline breathing which score "0" and on the other end "I can't breathe at all", which score "100" represent the worst difficulty perceived by patients.
Partial Pressure of Arterial Carbon Dioxide level | 1 hour
  Partial Pressure of Arterial Carbon Dioxide level change post intervention.
Rate of Intubation | 1 hour
  Intubation rate post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Adi Osman, Principal Investigator — Emergency Department, Hospital Raja Permaisuri Bainun

IPD SHARING:
Plan to Share IPD: No